CLINICAL TRIAL: NCT06484400
Title: Comparison of Cognitive Behavioral Therapy and Ericksonian Hypnosis Therapy for Depression and Anxiety Symptoms; Controlled Randomized Study
Brief Title: Cognitive Behavioral Therapy Versus Ericksonian Hypnosis Therapy for Depression and Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Asistant Professor, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nisantasi University
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Depression, Anxiety
Keywords: Cognitive Behavioral Therapy (CBT); Ericksonian Hypnotherapy; Depressive Disorder; Anxiety Disorders; Non-clinical Symptomatic Population
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Model Description: This study employs a randomized, controlled, parallel-group design to compare the effectiveness of Cognitive Behavioral Therapy (CBT) and Ericksonian Hypnotherapy in treating symptoms of depression and anxiety. The study includes three arms:
  CBT Group: Participants in this group will receive Cognitive Behavioral Therapy aimed at modifying negative thought patterns and behaviors to alleviate symptoms of depression and anxiety.
  Ericksonian Hypnotherapy Group: This group will undergo Ericksonian Hypnotherapy, which uses hypnosis and indirect suggestion to influence subconscious processes and mitigate psychological distress.
  Control Group: Participants in this group will not receive any intervention during the study period but will be monitored and offered therapy sessions after the study concludes, serving as a comparator to evaluate the efficacy of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy (CBT) Group (Experimental): Participants in this group will receive Cognitive Behavioral Therapy, which involves identifying and modifying negative thought patterns and behaviors to alleviate symptoms of depression and anxiety. Therapy sessions are conducted in person and on a one-on-one basis, ensuring tailored and direct therapeutic engagement. Each participant will attend 12 weekly sessions, each lasting approximately one hour.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Ericksonian Hypnotherapy Group (Experimental): This group will receive Ericksonian Hypnotherapy, a therapeutic approach that utilizes techniques of hypnosis and suggestion to access and alter subconscious processes, aiming to reduce psychological distress associated with depression and anxiety. Similar to the CBT group, sessions are delivered in person on a one-on-one basis, with a total of 12 weekly sessions, each one hour long.
  Interventions: Behavioral: Ericksonian Hypnotehrapy
- Control Group (No Intervention): Participants in this group will not receive any active intervention during the study period. This group serves as a control to measure the natural progression of depression and anxiety symptoms without therapeutic intervention. Participants will be monitored throughout the study and will be offered therapeutic sessions after the study's conclusion as compensation for their participation.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) is a well-established psychological treatment that focuses on identifying, understanding, and changing negative thinking and behavior patterns. The intervention involves structured sessions where participants are taught strategies to alter detrimental thoughts and behaviors to improve emotional regulation and develop personal coping strategies that target solving current problems. In this study, CBT will be delivered in 12 one-hour weekly sessions conducted in person and on a one-on-one basis. This intervention is designed to reduce symptoms of depression and anxiety through cognitive restructuring and behavioral adaptations.
  Arms: Cognitive Behavioral Therapy (CBT) Group
Behavioral: Ericksonian Hypnotehrapy — Ericksonian Hypnotherapy is a form of psychotherapy using clinical hypnosis and indirect suggestion to modify unconscious behaviors and thought patterns. Named after Dr. Milton H. Erickson, this therapeutic approach emphasizes adaptability and utilizes the patient's own experiences and internal resources for healing. The therapy is known for its effectiveness in addressing anxiety and depression by encouraging flexibility in perception and behavior. Like CBT, this intervention will be administered over 12 one-hour sessions, each conducted in person and tailored to the individual's unique psychological landscape.
  Arms: Ericksonian Hypnotherapy Group

SUMMARY:
Title: Comparison of Cognitive Behavioral Therapy and Ericksonian Hypnosis Therapy for Depression and Anxiety Symptoms; A Controlled Randomized Study.

Principal Investigator: Dr. Metin Çınaroğlu, Istanbul Nişantaşı University, Department of Psychology.

Study Duration: October, 2023 - Ongoing.

Objective: The study aims to compare the effectiveness of Cognitive Behavioral Therapy (CBT) and Ericksonian Hypnotherapy in alleviating symptoms of depression and anxiety among volunteers in Istanbul.

Methods: This randomized controlled trial will enroll healthy individuals aged 18-65 who exhibit symptoms of depression and anxiety but are not clinically diagnosed. Participants will be randomly divided into three groups: one receiving CBT, another receiving Ericksonian Hypnotherapy, and a control group receiving no therapeutic intervention. Standard psychological assessment tools such as the Beck Depression Inventory and Beck Anxiety Inventory will be used to measure outcomes.

Significance: Depression and anxiety are prevalent psychological disorders that significantly impair quality of life. Comparing these two therapeutic approaches may provide valuable insights into more effective psychological treatment strategies, thereby enhancing patient care in mental health settings.

Study Protocol:

Recruitment: 150 volunteers will be screened using socio-demographic forms and psychological assessments.

Intervention: Participants will undergo CBT or Ericksonian Hypnotherapy according to their group allocation, while the control group will be observed without intervention.

Evaluation: Pre- and post-treatment assessments will gauge the therapy's impact on depression and anxiety symptoms.

Expected Outcome: The study expects to demonstrate the relative efficacy of CBT and Ericksonian Hypnotherapy, providing evidence to guide treatment choices for managing depression and anxiety symptoms.

DETAILED DESCRIPTION:
Study Title: Comparison of Cognitive Behavioral Therapy and Ericksonian Hypnosis Therapy for Depression and Anxiety Symptoms; A Controlled Randomized Study.

Principal Investigator: Dr. Metin Çınaroğlu, Associate Professor, Department of Psychology, Istanbul Nişantaşı University.

Co-Investigators:

Expert Psychologist Dr. Eda Yılmazer, Department of Psychology, Beykoz University.

Psychologist Cemre Odabaşı, Clinical Psychology (Thesis) Student, Istanbul Nişantaşı University.

Dr. Selami Varol Ülker, Department of Psychology, Üsküdar University. Prof. Dr. Gökben Hızlı Sayar, Psychiatrist, Department of Psychiatry, Üsküdar University.

Study Duration: Start Date: October, 2023 - End Date: Ongoing.

Background and Rationale: Depression and anxiety are common mental health conditions globally, significantly impacting individuals' quality of life. Cognitive Behavioral Therapy (CBT) is widely recognized for its effectiveness in modifying dysfunctional thinking and behaviors associated with psychological disorders. Ericksonian Hypnotherapy, utilizing hypnotic suggestion and accessing unconscious processes, offers a complementary approach. This study aims to evaluate and compare the therapeutic efficacy of these interventions in non-clinically diagnosed, yet symptomatic individuals.

Objective: To compare the effectiveness of Cognitive Behavioral Therapy and Ericksonian Hypnotherapy in reducing symptoms of depression and anxiety.

Study Design: This is a randomized, controlled, comparative trial involving three groups:

CBT group (15 participants) Ericksonian Hypnotherapy group (15 participants) Waiting list control group (15 participants)

Methods:

Participants: A total of 150 volunteers from Istanbul, aged 18-65, displaying symptoms of depression and anxiety without a clinical diagnosis. Screening will be conducted using socio-demographic forms, the Beck Depression Inventory (BDI), and the Beck Anxiety Inventory (BAI).

Intervention: Participants will be randomly assigned to receive either CBT or Ericksonian Hypnotherapy, with each intervention being administered over 12 sessions. Each session will be conducted in person and on a one-on-one basis, lasting approximately one hour, held once a week.

Control Group: Individuals in the control group will not receive any intervention during the study period but will be offered therapy sessions after the study's conclusion as compensation for their participation.

Measurements: Psychological assessments will be conducted at baseline and post-intervention using the BDI and BAI to measure changes in depression and anxiety symptoms.

Data Analysis: The effectiveness of the interventions will be analyzed using independent and paired t-tests to compare pre- and post-intervention scores within and between groups. ANOVA will be utilized for comparing the three groups, and effect sizes will be calculated to determine the clinical significance of the treatments.

Ethical Considerations: The study will adhere to the ethical standards of the Helsinki Declaration and has been approved by the Institutional Review Board of Istanbul Nişantaşı University numbered 2023/3. Informed consent will be obtained from all participants, ensuring confidentiality and the right to withdraw from the study at any time without any consequences.

Significance: By directly comparing two distinct therapeutic modalities, this study seeks to provide empirical evidence to inform clinical practices and potentially guide future psychological interventions aimed at treating depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 18 and 65 years old.
* Symptoms: Participants must display symptoms of depression and/or anxiety, but not necessarily have a clinical diagnosis.
* Voluntary Participation: Participants must voluntarily agree to participate and must be able to provide informed consent.
* Residency: Participants must reside in or near the study location (Istanbul) to attend in-person sessions.
* Language: Participants must be proficient in the language in which the therapy is delivered (presumably Turkish).
* Availability: Participants must be available to attend all scheduled sessions over the course of the study (12 weekly sessions).

Exclusion Criteria:

* Psychiatric Diagnosis: Individuals with a severe psychiatric disorder requiring immediate or intensive intervention (e.g., schizophrenia, bipolar disorder, or severe depression with suicidal ideation).
* Current Psychotherapy: Individuals currently receiving other forms of psychotherapy or psychological treatment.
* Substance Abuse: Individuals with active substance abuse issues or dependencies that could interfere with therapy.
* Cognitive Impairments: Individuals with cognitive impairments or neurological disorders that would limit their ability to participate fully in therapy.
* Medical Conditions: Individuals with severe medical conditions that could interfere with participation in the study or pose a risk during the therapy sessions.
* Language Barrier: Non-Turkish speakers or those who do not understand the language well enough to benefit from therapy conducted in Turkish.
* Previous Participation: Individuals who have previously participated in similar studies or interventions, to avoid potential biases in responses and outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory (BDI) Scores | Baseline and 12 weeks post-intervention
  This outcome measures the change in depression levels among participants, as assessed by the Beck Depression Inventory. The BDI is a 21-item self-reported inventory that rates the severity of depression symptoms such as sadness, pessimism, sense of failure, and satisfaction in life, among others. The primary measure will be the difference in scores from baseline (pre-intervention) to post-intervention, indicating the efficacy of Cognitive Behavioral Therapy and Ericksonian Hypnotherapy in reducing depressive symptoms.
Change in Beck Anxiety Inventory (BAI) Scores | Baseline and 12 weeks post-intervention
  This outcome measures the change in anxiety levels, assessed using the Beck Anxiety Inventory. The BAI is a 21-item self-reported scale that evaluates the severity of anxiety symptoms, including nervousness, fear, and physiological responses related to anxiety. The main focus will be on the difference in scores from baseline to after the completion of the interventions, showcasing the impact of the therapeutic approaches on anxiety reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Cemre Odabaşı, MA, Principal Investigator — Clinical Psychology MA Student; Fadime Çınar, phd, Principal Investigator — Associate Professor
Locations (1):
- Metin Çınaroğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Description: The research team intends to make de-identified individual participant data (IPD) and supplementary materials available to further scientific investigation, ensure transparency, and encourage data reuse.
  Data and Supplementary Materials to be Shared: The shared dataset will include de-identified demographic data, baseline and post-intervention outcomes measured by the Beck Depression Inventory and the Beck Anxiety Inventory, session attendance records, and any additional assessments performed as part of the study. Supplementary materials such as session protocols, statistical analysis scripts, and intervention manuals will also be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The dataset and supplementary materials will be available indefinitely to maximize the impact and utility of the research contributions.
Access Criteria: All materials will be accessible without the need for a specific request or proposal submission, promoting an open and collaborative research environment.
URL: http://figshare.com